## Study Protocol

## Inclusion Criteria:

- 1. To be between the ages of 18-50,
- 2. Volunteering to participate in the research,
- 3. Those who have done aerobic exercise at least three days a week in the last three months

## Exclusion Criteria:

- 1. Neurological deficits in the upper or lower extremities,
- 2. Fractures or orthopedic problems in the upper or lower extremities,
- 3. Cardiovascular diseases that prevent rehabilitation,
- 4. Systematic rheumatic disease (rheumatoid arthritis, ankylosing spondylitis),
- 5. History of surgery in the last three months,
- 6. Patients with spine problems,
- 7. Smokers,
- 8. Patients with chronic respiratory problems.

Passed COVID-19 (n=25)

COVID-19 Proof (n=25)

- 1.Pulmonary Function Test
- 2. Respiratory Muscle Strength
- 3.Six Minute Walk Test (6MWT)
- 4.McGill Core Endurance Test
- 5. International Physical Activity Questionnaire Short Form (IPAQ-SF)
- 6. Quality of Life Scale (SF36)
- 7. Dyspnea Scale